CLINICAL TRIAL: NCT00991965
Title: An Open Label, Non-randomized, Single-arm, Multi-center Study to Assess Localized Alveolar Ridge Augmentation Utilizing INFUSE® Bone Graft Concurrent With Dental Implant Placement
Brief Title: Localized Alveolar Ridge Augmentation With Dental Implant
Acronym: RidgeDI
Status: Terminated | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Collaborators: Averion International Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: P09-03
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2011-10

CONDITIONS: Alveolar Bone Loss
Keywords: Alveolar Ridge Augmentation; Dental Implantation, Endosseous; Osseointegration; Bone Morphogenetic Proteins
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INFUSE® Bone Graft: all study participants will receive INFUSE® Bone Graft
  Interventions: Device: INFUSE® Bone Graft

INTERVENTIONS:
Device: INFUSE® Bone Graft — Patients will be treated with the commercially available INFUSE® Bone Graft material applied to an ACS in the area of the dental implant on Day 0 (Surgery). A follow-up visit will take place 2 weeks after implant of the INFUSE® Bone Graft material, or as regularly scheduled as per the standard of care (SOC) for the facility. Patients will return to the facility for final End of Study (EOS) assessments 6 months after surgery for placement of the appropriate prosthetic, and assessment of osseointegration and stability. Between the follow-up visit and the EOS visit, patients will be seen as per the SOC schedule for the facility.

SUMMARY:
The purpose of this research study is to shorten the treatment time course for patients who are scheduled for surgery to have a dental implant(s) placed into the upper front part of their mouths and need to have more bone in their jaws to support the implant.

DETAILED DESCRIPTION:
The INFUSE® Bone Graft is a device approved by the FDA to be used instead of using your own bone (from another site on your body) to replace missing bone in your jaw. INFUSE® Bone Graft is commercially available and is made up of 2 parts - recombinant human Bone Morphogenetic Protein-2 (rhBMP 2) placed on an absorbable collagen sponge (ACS). The rhBMP-2 is a genetically altered protein which recruits bone-forming cells to the surgical area and changes local cells to bone. ACS is made from Type I collagen from bovine (cattle) tendon. It helps to hold the rhBMP-2 in place and acts as a support for the growing bone. The sponge itself will reabsorb in time as the new bone forms.

The purpose of this research study is to shorten the treatment time course for the patients. This post-market study has been designed to further evaluate the effectiveness and safety of INFUSE® Bone Graft, along with dental implant placement, in a single procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. ≥18 years
3. Scheduled for dental implant into maxillary alveolar ridge
4. Negative urine pregnancy test for patients of child bearing potential and agreement not become pregnant for at least 12 months after surgery
5. Is able to comply with all study-related procedures, including exercising good oral hygiene
6. A prosthodontic treatment plan has been drafted.

Exclusion Criteria:

1. Known hypersensitivity to rhBMP-2, bovine Type I collagen or other components of the formulation
2. Known hypersensitivity to titanium
3. Operative site is in the area of a resected or extant tumor
4. Any active malignancy or current treatment for a malignancy
5. Active infection at operative site
6. History of prior exposure to rhBMP-2/ACS
7. Received and failed a previous alveolar ridge augmentation procedure
8. Pathology that would either compromise a bone grafting procedure, or interfere with obtaining quantitative measurements from postoperative CT scans
9. Significant untreated periodontal disease (> Grade III), caries, or chronic inflammation of the oral cavity at operative site
10. Active use of any nicotine-containing products such as, but not limited to, smoking and chewing tobacco, nicotine patch, nicotine gum, etc.
11. Insulin-dependent diabetic, or has known HgbA1c levels >6.5 %
12. History of malignancy within the past 5 years except for basal cell or squamous cell carcinoma of the skin
13. Patients who are lactating
14. History of metabolic bone disease, excluding idiopathic osteoporosis
15. History of autoimmune disease (e.g., documented multiple allergies, systemic lupus erythematosus, dermatomyositis, etc.) or immunosuppressive disease (e.g., Human Immunodeficiency Virus or Acquired Immune Deficiency Syndrome)
16. History of immune deficiency due to other treatments (e.g., radiation therapy, chemotherapy, steroid therapy)
17. History of adverse reaction to prior exposure to silicone or injectable collagen
18. Treatment with an investigational therapy within 1 month before the surgical procedure or plans to be treated with an investigational therapy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing bone augmentation of the alveolar ridge prior to placement of dental implants
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Stability and osseointegration of endosseous dental implants | 6 months post-implantation

SECONDARY OUTCOMES:
Evaluate evidence of successful initial INFUSE® Bone Graft and dental implant placement. Assess percent bone fill within the defect and safety of INFUSE®. Outcomes will be assessed via CT scans and periapical X-rays. | 6 months post-implantation

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Loma Linda, California
  - Los Angeles, California
  - Sarasota, Florida
  - Denver, North Carolina
  - Portland, Oregon
  - San Antonio, Texas